CLINICAL TRIAL: NCT04282499
Title: Comparative Effects of 12-weeks of Aerobic Versus Combined Exercise Training on Short Term Blood Pressure Variability in Patients With Hypertension
Brief Title: Effects of Exercise Training on Blood Pressure Variability
Acronym: VARIABILITA'
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele Roma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RP 24/18
Record Dates: First submitted 2020-02-17; First posted 2020-02-24 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2020-02

CONDITIONS: Hypertension; Cardiac Disease
Keywords: Hypertension; Cardiac Disease; Excercise
MeSH Terms: conditions — Hypertension; Heart Diseases | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: clinical evaluating the effects of 2 exercise training modalities on blood pressure variability. Recruited subjects will be randomized in two interventional arms: 1) aerobic exercise; 2) combined exercise (aerobic+resistance training).
Who Masked: Participant
Masking Description: Patients are not aware to the study design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combined exercise (Experimental): combined exercise (aerobic+resistance training)
  Interventions: Procedure: combined exercise
- aerobic exercise (Active Comparator): aerobic exercise only
  Interventions: Procedure: aerobic exercise

INTERVENTIONS:
Procedure: combined exercise — Patients will be undergone to aerobic exercises in addition to the resistance training.
  Arms: combined exercise
Procedure: aerobic exercise — Patients will be trained through the aerobic exercises only.
  Arms: aerobic exercise

SUMMARY:
A Randomized clinical evaluation of the effects of 2 exercise training modalities on blood pressure variability. Recruited subjects will be randomized in two interventional arms: 1) aerobic exercise; 2) combined exercise (aerobic+resistance training).

DETAILED DESCRIPTION:
This study will be a randomized trial, with two intervention arms: 1) Aerobic training (AT) and 2) Combined training (CT) groups. The planned training period will be 12 weeks for each group. Patients of both groups will be asked to exercise three times a week. Each session will last 80 minutes for each group. Population: We will includ 60 male subjects ≥ 45 years old, with established diagnosis of hypertension (of at least one year), treated with pharmacological therapy and with resting BP values under acceptable control (systolic BP <150 mmHg; diastolic BP < 90 mmHg) at admission. All groups of anti-hypertensive drugs will be admitted; there will be no restriction on the number of anti-hypertensive drugs taken by the patients. Sustained BP increase during the exercise protocol will be managed with the administration of furosemide (25-50 mg/daily). Patients who will need further pharmacological interventions for lowering BP will be withdrawn from the study. The following exclusion criteria will be adopted: secondary hypertension; significant heart valve diseases; signs and or symptoms of myocardial ischemia during ergometric test; neurological and or orthopedic conditions contraindicating or limiting ET; significant COPD (FEV1 <50%), or symptomatic peripheral arterial occlusive disease. Patients will be randomly assigned on 1:1 basis to either AT or CT group. The randomization code will be developed with a computer random-number generator to select random permuted blocks.

Exercise training protocols: AT group: every exercise session will include 10 min of warm-up, cool-down and flexibility exercises and 60 min of aerobic exercise with cycling and treadmill at 60-70% of VO2 peak.

CT group: patients will perform aerobic and resistance exercises in the same session. In order to balance the total amount of exercise, exercise sessions of the CT group will be organized as follow: 40 minutes of aerobic training with cycling and treadmill at 60-70% of VO2 peak; 20 minutes of resistance training including the following exercises: leg press and extension, shoulder press, chest press, low row and vertical traction. all the subjects Each strength exercise will be performed by patients at 60% of their maximal voluntary contraction. Patients of CT group will performed also 10 min of warm-up, cool-down and flexibility exercises. The one maximum repetition test (1RM) will be used to determine the RE load.

ELIGIBILITY:
Inclusion Criteria:

* ability to understand the study protocol instructions
* ability to sign the informed consent

Exclusion Criteria:

* sever cardio-vascular condition
* cognitive deficit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Change in 24/h systolic blood pressure variability | At baseline (day 1-T1) and at the end (12 weeks-T2) of the treatment.
  Systolic BP variability will be calculated through the formula of average real variability. This formula will be applied to the measures of BP obtained during 24 ambulatory BP monitoring

SECONDARY OUTCOMES:
Change in 24/h systolic and diatolic blood pressure values | At baseline (day 1-T1) and at the end (12 weeks-T2) of the treatment.
  Measures of BP obtained during 24 ambulatory BP monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Caminiti, MD, Principal Investigator — IRCCS San Raffaele Roma
Locations (1):
- IRCCS San Raffaele Pisana, Rome, RM, Italy